CLINICAL TRIAL: NCT06916195
Title: CMV PED Study - A Retrospective Observational Study To Understand The Clinical And Economic Burden Associated With Cytomegalovirus Reactivation and Related Health Outcomes In Pediatric Patients Receiving Allogeneic Hematopoietic Stem Cell Transplantation In Italy
Brief Title: Burden of Cytomegalovirus Reactivation in Pediatric Patients After Allogeneic Hematopoietic Stem Cell Transplantation
Acronym: CMV PED
Status: Recruiting | Type: Observational
Sponsor: MSD Italia S.r.l. (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS103043
Record Dates: First submitted 2025-03-31; First posted 2025-04-08 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-05

CONDITIONS: Cytomegalovirus Infection; Hematopoietic Stem Cells Transplantation
MeSH Terms: conditions — Cytomegalovirus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This observational retrospective analysis will provide useful information for clinicians and payers, and local guidelines committee members, to improve the understanding of Cytomegalovirus clinical and economic burden and clinical management of pediatric patients undergoing allogeneic Hematopoietic Stem Cells Transplantation in Italy.

DETAILED DESCRIPTION:
This is an observational retrospective analysis from the main pediatric centers in Italy (approximately 5 sites). The selected sites will be the most representative of Italy because they perform about 2/3 of all allogeneic HSCT per year.

Index date: date of allogeneic HSCT; retrospective data will be captured in consecutive patients undergoing allogeneic HSCT from January 2018 to June 2020 with maximum 12 months of follow-up for each patient. The data of the patients undergoing allogeneic HSCT after June 2020 will not be captured in order to avoid any possible bias due to off-label access to letermovir.

Medical Records (MR) will be used to describe the risk factors, patient characteristics, treatment patterns, and healthcare resource utilization of subjects who had a CMV infection.

Electronic or paper hospital charts (inpatient), clinical charts (inpatient and outpatient), and outpatient records will all be considered as MR for study purposes.

This is a secondary data collection study from electronic or paper medical chart review, no data from registry will be collected.

Patients (or their legally acceptable representatives) must have signed and dated the Informed Consent & Privacy Form (ICF), if applicable.

ELIGIBILITY:
Inclusion Criteria:

* Patients from birth to less than 18 years of age (at the moment of the allogeneic HSCT);
* Patients who received allogeneic HSCT between January 2018 and June 2020;
* Patients (or their legally acceptable representatives) must have signed and dated the Informed Consent & Privacy Form (ICF), if applicable.

Exclusion Criteria:

* Letermovir use at any time

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: About 230 patients from birth to less than 18 years of age allogeneic HSCT recipients at risk of developing CMV infection and/or disease who underwent allogeneic HSCT between January 2018 and June 2020 in the participating hospitals will be enrolled in the study. The selected hospitals will be the main ones in Italy based on the number of transplants performed every year and also considering the geographical distribution.
Sampling Method: Non-Probability Sample
Enrollment: 230 (Estimated)
Dates: Start 2025-05-09 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Summary of demographic and baseline characteristics | at baseline (day of transplant)
  Description through frequencies and percentages (for categorical variables) and mean and median values, SD, quartiles, interquartile ranges and extreme values (for continuous variables).
CMV Seroprevalence in the under 18 population undergoing allogeneic HSCT | at baseline (day of transplant)
  Proportion of patients CMV R+ at transplantation. CMV-seroprevalence and serostatus will be described according to the recipient or donor positivity. Comparisons will be conducted using the Chi-square or Fisher's exact test (for categorical variables), or the t-test or Wilcoxon rank sum test (for continuous variables).
CMV serostatus | at baseline (day of transplant)
  R+/D-, R+/D+ and R-/D+ combination frequencies. CMV-seroprevalence and serostatus will be described according to the recipient or donor positivity. Comparisons will be conducted using the Chi-square or Fisher's exact test (for categorical variables), or the t-test or Wilcoxon rank sum test (for continuous variables).
Donor type | at baseline (day of transplant)
  Allogeneic HSCT characteristics
Stem cell source | at baseline (day of transplant)
  Allogeneic Hematopoietic Stem Cells Transplantation characteristics
Conditioning intensity | at baseline (day of transplant)
  Allogeneic Hematopoietic Stem Cells Transplantation characteristics
Underlying condition | at baseline (day of transplant)
  Allogeneic Hematopoietic Stem Cells Transplantation characteristics
Usage of immunosuppression | at baseline (day of transplant)
  Allogeneic Hematopoietic Stem Cells Transplantation characteristics
Current standard of care in CMV management in terms of PET approach | during the first-year post-transplant
  It will be described quantitatively by tabulating frequencies and percentages.
Current standard of care in CMV management in terms of GCV prophylaxis | during the first-year post-transplant
  It will be described quantitatively by tabulating frequencies and percentages.
Current standard of care in CMV management in terms of ACV prophylaxis | during the first-year post-transplant
  It will be described quantitatively by tabulating frequencies and percentages.
Current standard of care in CMV management in terms of other | during the first-year post-transplant
  It will be described quantitatively by tabulating frequencies and percentages.

SECONDARY OUTCOMES:
Rate of clinically significant CMV infection | at day +100, day +200 and during the first year post allogeneic HCT
  Incidence rates will be computed by dividing the number of events by the total number of person-years and then multiplying per 100. A Kaplan-Meier curve will describe the timing of first CS-CMVi and mortality.
Median time to first CS-CMVi | during the first year after transplantation
  A Kaplan-Meier curve will describe the timing of first CS-CMVi and mortality.
Rate of viral infections other than CMV | at day +100, day +200 and during the first year post allogeneic HCT
  Incidence rates will be computed by dividing the number of events by the total number of person-years and then multiplying per 100. A Kaplan-Meier curve will describe the timing of first CS-CMVi and mortality.
Rate of bacterial infections | at day +100, day +200 and during the first year post allogeneic HCT
  Incidence rates will be computed by dividing the number of events by the total number of person-years and then multiplying per 100. A Kaplan-Meier curve will describe the timing of first CS-CMVi and mortality.
Rate of fungal infections | at day +100, day +200 and during the first year post allogeneic HCT
  Incidence rates will be computed by dividing the number of events by the total number of person-years and then multiplying per 100. A Kaplan-Meier curve will describe the timing of first CS-CMVi and mortality.
Allogeneic HSCT risk factors | at baseline (day of transplant)
  Underlying condition, donor type, stem cell source, conditioning intensity, immunosuppressive therapies.
  The relation between complications and risk factors will be analyzed through Cox regression models.
CMV-related complications | during the first-year post-transplant
  Proportion of patients with at least one CMV disease, "overall" and by type of disease, and number of diseases per patient.
  The relation between complications and risk factors will be analyzed through Cox regression models.
CMV-related complications | at day +100, day +200 and during the first year post allogeneic HCT
  Rate of acute and chronic Graft vs Host Disease Incidence rates will be computed by dividing the number of events by the total number of person-years and then multiplying per 100. A Kaplan-Meier curve will describe the timing of first CS-CMVi and mortality.
CMV-related complications | during the first-year post-transplant
  Rate of opportunistic infection declared by the investigator "CMV related-complication"
Number of hospitalizations and length of stay (LOS) after allogeneic HSCT | at day +100, day +200 and during the first year post allogeneic HCT
  Utilization of several healthcare resources will be described to quantify the economic burden. Data will include frequency of re-hospitalization, exams, diagnostic tests, visits, drugs use and the duration of re-hospitalization. Statistical tests (Chi-square, Fisher's exact, Student's T or Wilcoxon rank-sum) will be applied based on the variable type.
All-cause mortality rate | at day +100, day +200 and during the first year post allogeneic HCT
  Kaplan-Meier curves will describe the timing of events.

CONTACTS AND LOCATIONS:
Locations (5):
- Italy (5):
  - IRCCS Istituto Giannina Gaslini, Trapianto di Cellule Staminali Emopoietiche, Dipartimento di Onco-Ematologia Pediatrica, Genova
  - Ospedale San Gerardo, Clinica Pediatrica, Monza
  - Azienda Ospedale-Università di Padova, Clinica di Oncoematologia Pediatrica, Padua
  - IRCCS Ospedale Pediatrico Bambino Gesù, Dipartimento di Pediatria Ematologia e Oncologia, Roma
  - Ospedale Infantile Regina Margherita, Dipartimento Patologia e Cura del Bambino, Torino